CLINICAL TRIAL: NCT01808378
Title: Phase IIa Clinical Trial to Study the Feasability and Security of the Expanded Autologous Stem Cells (ASC) From Lipoaspirate in the Bilateral Limbic Associated Keratopathy Treatment
Brief Title: Stem Cells Treatment for Bilateral Limbic Associated Keratopathy (HULPOFT)
Acronym: HULPOFT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HULPOFT-2010-01; 2010-024328-53 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2012-09

CONDITIONS: Keratopathy
Keywords: Bilateral limbic associated keratopathy; Expanded Adipose Derived Stem Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Stem Cells (Experimental): Autologous expanded adipose-derived stem cells
  Interventions: Drug: Expanded adipose-derived stem cells

INTERVENTIONS:
Drug: Expanded adipose-derived stem cells — Local injection of autologousadipose derived stem cells
  Other Names: ASC

SUMMARY:
Evaluate the use of the autologous ASC for the treatment of bilateral limbic associated keratopathy

DETAILED DESCRIPTION:
Intralesional use by inject of adipose derived stem cells

ELIGIBILITY:
Inclusion Criteria:

1. -Signed informed consent
2. -Previously diagnosed bilateral limbic obstruction
3. -Men and women over 18 years old. Good general state of health according to the findings of the clinical history and the physical examination
4. -Suffering chronic keratopathy accomplishing the following criteria:

   * Confirmed limbic obstruction with an impression cytology
   * Repeated usual treatment failure for this pathology

Exclusion Criteria:

1. -Having suffered a neoplasia in the previous 5 years
2. -Local anesthesia allergies
3. -Patients having participate in any other study in the previous 90 days to the inclusion
4. -Patients on medication with tacrolimus or cyclosporine in the 4 previous week to the cellular therapy
5. -Any medical or psychiatric illness that, in the investigator opinion, could suppose a reason for the study exclusion
6. -Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from study
7. -Patients with congenital or acquired immunodeficiencies. HIV, HBV, HCV or treponema infection, whether active or latent
8. -Patients who have suffering major surgery or severe trauma in the prior 6 months
9. -Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the practicability and security of the autologous expanded lipoaspirated stem cells for the treatment of bilateral limbic associated keratopathy | 16 weeks
  Micro ocular Photography Visual acuity

SECONDARY OUTCOMES:
Quality of life assessment using the SF-12 Questionnaire | 1, 4, 16, 24 weeks
  SF-12 questionnaire
Adverse events | 1, 4, 16, 24 weeks
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: Ana Boto de los Bueis, MD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Nishida K. Tissue engineering of the cornea. Cornea. 2003 Oct;22(7 Suppl):S28-34. doi: 10.1097/00003226-200310001-00005. PMID 14703705
- [Background] Arntz Bustos A, Durán de la Colina JA. Anatomía funcional de la superficie ocular. En; Superficie Ocular. Ed S.E.O. 2004; 1-12
- [Background] Schermer A, Galvin S, Sun TT. Differentiation-related expression of a major 64K corneal keratin in vivo and in culture suggests limbal location of corneal epithelial stem cells. J Cell Biol. 1986 Jul;103(1):49-62. doi: 10.1083/jcb.103.1.49. PMID 2424919
- [Background] Tseng SC. Staging of conjunctival squamous metaplasia by impression cytology. Ophthalmology. 1985 Jun;92(6):728-33. doi: 10.1016/s0161-6420(85)33967-2. PMID 3897935
- [Background] Kenyon KR, Tseng SC. Limbal autograft transplantation for ocular surface disorders. Ophthalmology. 1989 May;96(5):709-22; discussion 722-3. doi: 10.1016/s0161-6420(89)32833-8. PMID 2748125
- [Background] Santos MS, Gomes JA, Hofling-Lima AL, Rizzo LV, Romano AC, Belfort R Jr. Survival analysis of conjunctival limbal grafts and amniotic membrane transplantation in eyes with total limbal stem cell deficiency. Am J Ophthalmol. 2005 Aug;140(2):223-30. doi: 10.1016/j.ajo.2005.03.022. PMID 16023069
- [Background] Chen JJ, Tseng SC. Corneal epithelial wound healing in partial limbal deficiency. Invest Ophthalmol Vis Sci. 1990 Jul;31(7):1301-14. PMID 1694836
- [Background] Tan DT, Ficker LA, Buckley RJ. Limbal transplantation. Ophthalmology. 1996 Jan;103(1):29-36. doi: 10.1016/s0161-6420(96)30737-9. PMID 8628556
- [Background] Samson CM, Nduaguba C, Baltatzis S, Foster CS. Limbal stem cell transplantation in chronic inflammatory eye disease. Ophthalmology. 2002 May;109(5):862-8. doi: 10.1016/s0161-6420(02)00994-6. PMID 11986089
- [Background] Tsubota K, Toda I, Saito H, Shinozaki N, Shimazaki J. Reconstruction of the corneal epithelium by limbal allograft transplantation for severe ocular surface disorders. Ophthalmology. 1995 Oct;102(10):1486-96. doi: 10.1016/s0161-6420(95)30841-x. PMID 9097796
- [Background] Ilari L, Daya SM. Long-term outcomes of keratolimbal allograft for the treatment of severe ocular surface disorders. Ophthalmology. 2002 Jul;109(7):1278-84. doi: 10.1016/s0161-6420(02)01081-3. PMID 12093650
- [Background] Pellegrini G, De Luca M, Arsenijevic Y. Towards therapeutic application of ocular stem cells. Semin Cell Dev Biol. 2007 Dec;18(6):805-18. doi: 10.1016/j.semcdb.2007.09.011. Epub 2007 Sep 16. PMID 17959397
- [Background] Inatomi T, Nakamura T, Koizumi N, Sotozono C, Yokoi N, Kinoshita S. Midterm results on ocular surface reconstruction using cultivated autologous oral mucosal epithelial transplantation. Am J Ophthalmol. 2006 Feb;141(2):267-275. doi: 10.1016/j.ajo.2005.09.003. PMID 16458679
- [Background] Yao YF, Inoue Y, Miyazaki D, Shimomura Y, Ohashi Y, Tano Y. Ocular resurfacing and alloepithelial rejection in a murine keratoepithelioplasty model. Invest Ophthalmol Vis Sci. 1995 Dec;36(13):2623-33. PMID 7499085
- [Background] Daya SM, Watson A, Sharpe JR, Giledi O, Rowe A, Martin R, James SE. Outcomes and DNA analysis of ex vivo expanded stem cell allograft for ocular surface reconstruction. Ophthalmology. 2005 Mar;112(3):470-7. doi: 10.1016/j.ophtha.2004.09.023. PMID 15745776
- [Background] Nakamura T, Kinoshita S. Ocular surface reconstruction using cultivated mucosal epithelial stem cells. Cornea. 2003 Oct;22(7 Suppl):S75-80. doi: 10.1097/00003226-200310001-00011. PMID 14703711
- [Background] Nakamura T, Inatomi T, Sotozono C, Amemiya T, Kanamura N, Kinoshita S. Transplantation of cultivated autologous oral mucosal epithelial cells in patients with severe ocular surface disorders. Br J Ophthalmol. 2004 Oct;88(10):1280-4. doi: 10.1136/bjo.2003.038497. PMID 15377551
- [Background] Nishida K, Yamato M, Hayashida Y, Watanabe K, Yamamoto K, Adachi E, Nagai S, Kikuchi A, Maeda N, Watanabe H, Okano T, Tano Y. Corneal reconstruction with tissue-engineered cell sheets composed of autologous oral mucosal epithelium. N Engl J Med. 2004 Sep 16;351(12):1187-96. doi: 10.1056/NEJMoa040455. PMID 15371576
- [Background] Lehrer MS, Sun TT, Lavker RM. Strategies of epithelial repair: modulation of stem cell and transit amplifying cell proliferation. J Cell Sci. 1998 Oct;111 ( Pt 19):2867-75. doi: 10.1242/jcs.111.19.2867. PMID 9730979
- [Background] Ma Y, Xu Y, Xiao Z, Yang W, Zhang C, Song E, Du Y, Li L. Reconstruction of chemically burned rat corneal surface by bone marrow-derived human mesenchymal stem cells. Stem Cells. 2006 Feb;24(2):315-21. doi: 10.1634/stemcells.2005-0046. Epub 2005 Aug 18. PMID 16109757
- [Background] Blazejewska EA, Schlotzer-Schrehardt U, Zenkel M, Bachmann B, Chankiewitz E, Jacobi C, Kruse FE. Corneal limbal microenvironment can induce transdifferentiation of hair follicle stem cells into corneal epithelial-like cells. Stem Cells. 2009 Mar;27(3):642-52. doi: 10.1634/stemcells.2008-0721. PMID 19074417
- [Background] Gu S, Xing C, Han J, Tso MO, Hong J. Differentiation of rabbit bone marrow mesenchymal stem cells into corneal epithelial cells in vivo and ex vivo. Mol Vis. 2009;15:99-107. Epub 2009 Jan 16. PMID 19156227
- [Background] Arnalich-Montiel F, Pastor S, Blazquez-Martinez A, Fernandez-Delgado J, Nistal M, Alio JL, De Miguel MP. Adipose-derived stem cells are a source for cell therapy of the corneal stroma. Stem Cells. 2008 Feb;26(2):570-9. doi: 10.1634/stemcells.2007-0653. Epub 2007 Dec 6. PMID 18065394
- [Derived] Boto de Los Bueis A, Vidal Arranz C, Del Hierro-Zarzuelo A, Diaz Valle D, Mendez Fernandez R, Gabarron Hermosilla MI, Benitez Del Castillo JM, Garcia-Arranz M. Long-Term Effects of Adipose-Derived Stem Cells for the Treatment of Bilateral Limbal Stem Cell Deficiency. Curr Eye Res. 2024 Apr;49(4):345-353. doi: 10.1080/02713683.2023.2297342. Epub 2023 Dec 28. PMID 38152876